CLINICAL TRIAL: NCT03668977
Title: Impact of a Balanced Protein-Energy Supplement in Pregnancy and Early Lactation on Reproductive Outcomes and Growth in Southern Nepal
Brief Title: Balanced Protein-Energy Supplement in Pregnancy and Early Lactation on Birth Outcomes and Growth in Southern Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Harvard University (Other); Johns Hopkins University (Other); Bill and Melinda Gates Foundation (Other); Thrasher Research Fund (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James M. Tielsch, PhD, Professor and Chair School of Public Health, PI, George Washington University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 081739
Record Dates: First submitted 2018-05-30; First posted 2018-09-13 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy and Early Lactation Among Women Living in an Area Endemic for Malnutrition

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Routine care (No Intervention): In all four groups, the following antenatal and post-natal interventions will be offered:
  * Women encouraged to enroll in routine antenatal care at their local health post/center.
  * A clean birthing kit consisting of a clean blade, string, and plastic disc for cutting the cord, a plastic sheet, a bar of soap, and a tube of chlorhexidine ointment for application to the umbilical stump.
  * Women encouraged to deliver at a certified birthing facility and participate in the government's incentive scheme.
  * Nutritional, hygiene, and infant care counseling.
  * Tetanus toxoid (if needed) and iron-folic acid supplements.
- Supplementation-pregnancy (Experimental): A daily fortified balanced protein-energy nutritional supplement beginning in the 2nd trimester and continuing throughout pregnancy. The exact form of this supplement will be selected in Phases one and two but its composition will be in conformance with the recommendations from the expert panel convened by the B&MGF on nutritional supplementation in pregnancy (Expert Consultation, 2016). The calorie content will be approximately 400 Kcal/day with approximately 14 g of protein.
  Interventions: Dietary Supplement: Fortified balanced protein-energy.
- Supplementation-lactation (Experimental): A daily fortified balanced protein-energy nutritional supplement beginning after delivery and continuing through 6 months post-partum. The exact form of this supplement will be selected in Phases one and two but its composition will be in conformance with the recommendations from the expert panel convened by the B&MGF on nutritional supplementation in pregnancy (Expert Consultation, 2016). The calorie content will be approximately 400 Kcal/day with approximately 14 g of protein.
  Interventions: Dietary Supplement: Fortified balanced protein-energy.
- Supplementation-pregnancy & lactation (Experimental): A daily fortified balanced protein-energy nutritional supplement beginning in the 2nd trimester and continuing through 6 months post-partum. The exact form of this supplement will be selected in Phases one and two but its composition will be in conformance with the recommendations from the expert panel convened by the B&MGF on nutritional supplementation in pregnancy (Expert Consultation, 2016). The calorie content will be approximately 400 Kcal/day with approximately 14 g of protein.
  Interventions: Dietary Supplement: Fortified balanced protein-energy.

INTERVENTIONS:
Dietary Supplement: Fortified balanced protein-energy. — The exact form of this supplement will be selected in Phases one and two but its composition will be in conformance with the recommendations from the expert panel convened by the B&MGF on nutritional supplementation in pregnancy (Expert Consultation, 2016). The calorie content will be approxmately 400 Kcal/day with approximately 14 g of protein.
  Arms: Supplementation-lactation; Supplementation-pregnancy; Supplementation-pregnancy & lactation

SUMMARY:
This project will test the efficacy of a balanced protein energy supplement for daily use during pregnancy and the first 6 months after delivery on the outcomes of pregnancy and growth of infants during the first 6 months of life. Approximately 1800 pregnant women from a district in southern Nepal will be recruited and randomly assigned to one of 4 groups, control in pregnancy & post-partum, supplementation in pregnancy & control post-partum, control in pregnancy & supplementation post-partum, or supplementation in pregnancy & post-partum. Pregnancies will be followed until delivery and the infants through 6 months of age. Outcomes of interest include birth size (weight and length), gestational age at delivery, maternal weight gain in pregnancy, maternal weight at 6 months post-partum, infant growth, and breast milk composition.

DETAILED DESCRIPTION:
Background Undernourished women in many low and middle income countries (LMICs) enter pregnancy with low nutritional reserves, and low maternal body mass index (BMI) and short stature are associated with increased risks of a variety of adverse reproductive outcomes (Kozuki et al., 2015; Rahman et al., 2015). Balanced protein-energy (BE-P) supplementation during pregnancy shows moderate evidence than such dietary supplementation can decrease the risk of stillbirth and small-for-gestational-age (SGA) births (Ota et al., 2015; Stevens et al., 2015). The WHO antenatal care guidelines recommend providing pregnant women in undernourished populations with balanced protein energy dietary supplementation (WHO, 2016). The current evidence base for BP-E supplementation draws from a number of studies where BP-E supplements varied widely in composition and form (Imad & Bhutta, 2002). Recent studies using fortified blended foods found that although approximately 800 kcal/d was provided, the net energy intake increased by a much smaller amount (200-300 kcal) (Janmohamed et al., 2016; Saville et al., unpublished trial in Nepal).

Evidence regarding dietary practices and preferences among pregnant women in Nepal is generally limited, however, some studies have shown that intra-household food allocation and specific food beliefs/behaviors do not favor adequate energy or micronutrient intake among adolescent girls and adult women (Gittelsohn, 1991; Gittelsohn et al., 1997). Christian et al showed that staple food intake can be reduced during pregnancy; which could be attributed to an aversion to food, lack of appetite, feeling unwell, or concern regarding having a "large" baby and difficulties with labor and delivery (Christian et al., 2006). Low nutrition knowledge may also play a role in suboptimal intake among women (Jones et al., 2005). Dynamic changes in access and use of services offer the opportunity to nest additional nutritional support services within the antenatal care system, including BP-E supplementation. However, information is limited regarding the impact such supplementation will have on the key birth outcomes that affect child health and development. It is this lack of evidence that this project will address.

Methods This project will be done in three phases. Phase one will identify preferable supplement types for use in pregnancy in the South Asian context. Phase two will use the results of phase one to conduct a medium-term feeding trial to assess acceptability and consumption. Phase three will be a large, community-based randomized trial using at least one of these supplement options for use in pregnancy and through the first 6 months post-partum on birth outcomes and early infant growth.

Specific Aim, Phase 1: Identify preferred product types for the provision of fortified BEP supplements among pregnant women in Southern Nepal.

Specific Aim, Phase 2: Assess the 8-week acceptability and consumption of 2 selected supplements with nutrient content consistent with Bill and Melinda Gates Foundation (BMGF) guidance among pregnant women in Southern Nepal.

Specific Aims Phase 3: Community-Based Randomized Field Trial

There is one primary aim and a number of secondary aims for each marginal treatment arm of this trial. Primary aims:

1. To compare the incidence of small-for-gestational-age (SGA) newborn infants born to mothers randomized to receive either a daily balanced protein-energy nutritional supplement with multiple micronutrients or control during pregnancy. SGA will be defined as <10th centile of birthweight for gestational age standard using InterGrowth 21st criteria (Villar et al., 2014).
2. To compare the growth of live-born infants among mothers randomized to the two groups during the first 6 months post-partum. The primary infant growth outcome is Length-for-Age Z (LAZ) score using the WHO Child Growth Study criteria (WHO, 2006).

Secondary aims:

Pregnancy Supplementation

1. To compare the incidence of short-for-gestational-age (ShGA) newborn infants born to mothers randomized to the two groups during pregnancy. ShGA defined as <10th centile of birth length for gestational age standard using InterGrowth 21st criteria.
2. To compare the incidence of small-for-gestational-age (SGA) newborn infants born to mothers randomized to the two groups during pregnancy. SGA defined as <3rd centile of birthweight for gestational age standard using InterGrowth 21st criteria.
3. To compare the incidence of short-for-gestational-age (ShGA) newborn infants born to mothers randomized to the two groups during pregnancy. ShGA defined as <3rd centile of birth length for gestational age standard using InterGrowth 21st criteria.
4. To compare the means and distribution of birth weight, birth length and gestational age (and percent <2500 gm, <37 weeks gestation) in infants born to women randomized to the two groups during pregnancy.
5. To compare the growth through 6 and 12 months of age (LAZ, weight-for-age Z (WAZ), weight-for-length Z (WLZ) scores) of infants born to women randomized to the two groups during pregnancy. 12 months follow-up will be available on approximately 2/3rd of infants.
6. To compare maternal weight gain during pregnancy among women randomized to the two groups during pregnancy.
7. To compare the diversity of the gut microbiome in pregnancy among women randomized to receive either a daily balanced protein-energy nutritional supplement with multiple micronutrients or control during pregnancy.

Post-Partum Supplementation

1. To compare WAZ and WLZ scores through 6 and 12 months of age of infants born to women randomized to receive either a daily balanced protein-energy nutritional supplement or control during the first 6 months post-partum. 12 months follow-up will be available on approximately 2/3rd of infants and women.
2. To compare the weight and BMI of mothers at 6 and 12 months post-partum among women randomized to the two groups during the first 6 months post-partum. 12 months follow-up will be available on approximately 2/3rd of mothers.
3. To compare the diversity of the gut microbiome post-partum among women randomized to receive either a daily balanced protein-energy nutritional supplement with multiple micronutrients or control during post-partum.
4. To compare the diversity of the gut microbiome among infants <6 months of age whose mothers were randomized to receive either a daily balanced protein-energy nutritional supplement or control during the post-partum period.
5. To compare the neurodevelopmental status of infants at 6 months of age whose mothers were randomized to receive either a daily balanced protein-energy nutritional supplement of control during the post-partum period.

Combination of Pregnancy and Post-Partum Supplementation

1. To compare the impact of combined pregnancy and post-partum nutritional supplementation with women who received only pregnancy or post-partum supplementation alone on LAZ, WAZ, and WLZ scores at 6 and 12 months of age among infants born to these mothers. 12 months follow-up will be available on approximately 2/3rd of infants.

Study Design for Phases 1 & 2: A two-phase, mixed methods approach combining qualitative and quantitative methods for data collection will be used.

Phase 1: 11 product types will be introduced to participants in a single-meal test for their feedback on acceptability. Phase 1 will collect data to describe general preferences across product types and variations.

Phase 2: 2 product types identified in Phase 1 will be tested in an 8-week feeding trial. Each participating woman will experience one selected product type for a total of 8 weeks. Hedonic properties will be assessed at 2 and 8 weeks.

Complementary qualitative data will also be collected using in-depth interviews and focus group discussions during both phases 1 and 2.

Setting for all Phases This project will be conducted in a chronically food insecure study site in southern Nepal (Sarlahi District). This site is representative of a region (South Asia) and meets the criteria of having adequate local security conditions and presence of a strong field research site.

Study population and sample size estimates Phases 1 & 2:

Pregnant Women (PW): In Phase 1, a convenience sample of 40 PW will be selected to evaluate 11 product types. In Phase 2, women participating in the home feeding trial (n = 40 for each of two product types, total n=80) will additionally participate in in-depth interviews.

Data Collection: Phases 1 & 2:

Phase 1. Identify preferred product types Direct observation of single meal with hedonic testing: During the single meal observation, each participant will receive 1 serving of each product. Acceptability will be assessed based on Likert-like scoring using hedonic scales of overall liking, appearance, smell, taste and consistency.

Focus group discussion: Focus groups (maximum of 40 women) will be conducted following the single meal direct observation.

Phase 2. Home-feeding trial to assess acceptability and at-home consumption Two product types selected in Phase 1 will be assessed for medium-term acceptability and utilization through an 8-week feeding trial. Two measures of adherence will be assessed at each weekly home distribution; adherence in the last 24 hours using direct questioning and adherence using direct sachet/packet count.

Hedonic testing: Hedonic testing will be done at 8 weeks (de Graaf et al., 2005).

In-depth interviews: For both products, interviews will be conducted with PW and other household members, and health staff.

Focus group discussions: Focus groups among PW receiving both products will be conducted at the end of Phase 2.

Data analysis, Phases 1 & 2:

Adherence data: Adherence by self-report will be calculated as the percentage of days the supplement was reported to be consumed and mean portion when consumed, and adherence by sachet count will be calculated as total empty packages returned divided by total packages expected to be consumed.

Hedonic test data: Product liking, and left over quantities over time will be summarized by product type using means for continuous variables.

Qualitative data: Analysis will be ongoing throughout data collection, and conducted by the research team using an exploratory, inductive approach that will draw from Grounded Theory and allow for the analysis of emergent themes (Charmaz, 2014; Ridder et al., 2014; Charmaz, 2006). Data will be systematically coded using Dedoose computer software (Consultants, 2016) (Glesne & Peshkin, 1992).

Phase 3: Randomized Trial Design The design of this study is a community-based, household level-randomized 2x2 factorial trial among women who become pregnant in the study area. Due to interruptions due to the COVID-19 pandemic and funding issues, recruitment was conducted in two non-concurrent cohorts with 50% of recruitment during each cohort.

Study Population The study population for this trial will include all women who become pregnant during two cohorts each over an approximate 6 month period in a set of Nagarpalikas or Gaunpalikas in Sarlahi District, Nepal. Newly pregnant women will be identified through a pregnancy surveillance system.

Intervention

Two interventions strategies will be tested in a factorial design in this trial; nutritional supplementation during pregnancy and nutritional supplementation during the first 6 months post-partum. The exact forms of this supplement will be selected in Phases one and two but its composition will be in conformance with the recommendations from the expert panel convened by the BMGF on nutritional supplementation in pregnancy (Expert Consultation, 2016). Women in households allocated to the control groups will receive a standard package of antenatal services and nutritional counseling by study staff. In all four groups, the following antenatal and post-natal interventions will be offered:

* Women will be encouraged to enroll in routine antenatal care at their local health post/center.
* A clean birthing kit will be provided consisting of a clean blade, string, and plastic disc for cutting the cord, a plastic sheet, a bar of soap, and a tube of chlorhexidine ointment for application to the umbilical stump.
* Women will be encouraged to deliver at a certified birthing facility and participate in the government's incentive scheme.
* Additional nutritional, hygiene, and infant care counseling will be provided by study staff.
* If a woman reports not attending ANC and/or not receiving tetanus toxoid or iron-folic acid supplements, our study staff will provide them.

Masking While it will not be possible to mask the participants or the Ward Data Collectors to the treatment assignment, we will attempt to mask the birth and growth assessment teams to the treatment assignments.

Randomization Randomization will be done at the household level for this study. This means that once the first pregnant woman from a given household is identified and consents to be in the trial, that household will be allocated to either the supplement or non-supplement group (for pregnancy). Any other woman or women from this household who subsequently become pregnant within the 9-month enrollment period, would also be assigned to that group.

We will pre-generate a randomization sequence denoting the two pregnancy allocation possibilities (supplement, no-supplement) using the R software environment for statistical programming (www.r-project.org) using randomly permuted blocks of size 4, 8, and 12, to ensure sequential balance across the groups throughout the enrollment period.

For randomization to the post-delivery exposure (i.e. supplement, no-supplement), a slightly modified procedure will be followed. Here, we will construct two pre-generated allocation sequences, again constructed with randomly permuted blocks of size 4, 8, and 12. These two sequences will be stored in our database, and annotated/labelled to allow for allocating post-delivery exposures stratified by pregnancy exposure.

Substudies A group of substudies will be conducted among a systematic sample of 120 pregnant women per treatment group (total of 240). These substudies include assessments of maternal dietary intake, the gut microbiome using multiplex PCR and metabolomic assays in stool, and infant neurodevelopmental outcomes at 6 months.

Maternal Microbiome SubStudy The objective is to examine whether a BP-E nutritional supplement during pregnancy and breastfeeding will promote a more diverse and normal gut microbiome in pregnant and breastfeeding women.

Methods:

Stool will be collected among all 120 women per group at the following times:

* at the time of baseline enrollment in early pregnancy.
* at the late pregnancy visit (~34 weeks gestation).

Dietary Intake Sub-Study The purpose of this sub-study is to assess whether there is significant dietary diversion occurring in the supplementation groups compared with controls. We will use daily energy and protein intake as the primary indicators of diversion. A quantitative 24-hour recall instrument will be used once in pregnancy (in duplicate) and once in the post-partum period (in duplicate). We will adapt dietary instruments that have been used previously in this population for this sub-study (Sudo et al, 2006; Parajuli et al, 2012; Campbell et al, 2014; Henjum et al, 2015).

Sample Size / Power Calculations These calculations assume the nutritional supplementation in pregnancy and post-partum periods have independent effects on the outcomes of interest. We are not powered to detect specific interaction effects on either primary or secondary outcomes.

Primary Outcomes: Small-for-gestational-age (SGA) is the primary outcome that we have used to drive the sample size calculations. While not a truly individually randomized trial (households will be randomized), the very small likelihood of identifying more than one eligible pregnant women in a household over a 9 month period is quite low (<3.5% of "clusters" will have more than 1 individual outcome). We've estimated the effect of this level of clustering on sample size and found it to be extremely small versus individual randomization. Therefore, all our sample size/power estimates are based on individual randomization.

Over a period of two phases of approximately 6 months, we expect that eligible households in our study area will yield approximately 1600 pregnant women whose infants will be seen within 72 hours of birth for measurement of the primary birth outcome.

Table: Effect Size Detectable for Primary Birth Outcome Given 774 Infants per Group Measured within 72 Hours of Birth Outcome Relative Risk Detectable (Supplemented/Unsupplemented) 80% Power 90% Power Primary SGA (10th centile) 0.825 0.798

We will be able to detect a 17.5% reduction in SGA with 80% power and a 20.2% reduction with 90% power assuming a type 1 error of 5% (two-sided).

The table below presents the detectable relative risks or mean differences for a variety of secondary outcomes with 80% and 90% power.

Table: Detectable Difference in Secondary Outcomes (Marginal Comparisons) Outcome Detectable Relative Risk or Difference Between Groups 80% Power 90% Power Secondary ShGA (10th centile)a 0.778 0.745 SGA (3rd centile)b 0.726 0.686 ShGA (3rd centile)c 0.653 0.604 Mean Birth Weight d 60.7 g 70.2 g Mean Birth Length e 3.0 mm 3.5 mm LAZ at 6 months1 0.16 Z scores 0.18 Z Scores WAZ at 6 months2 0.17 Z scores 0.20 Z scores WLZ at 6 months3 0.18 Z scores 0.21 Z scores Maternal Weight Gain in Pregnancy4 463 g 536 g Maternal Weight at 6 months Post-Partum5 0.89 kg 1.03 kg

a ShGA (10th centile expected rate is 30.1%. b SGA (3rd centile) expected rate is 22.1%. c ShGA (3rd centile) expected rate is 14.4%. d Expected mean birth weight is 2708 g (SD=429). e Expected mean birth length is 47.6 cm (SD=2.2).

1. Expected mean LAZ at 6 months is -1.04.
2. Expected mean WAZ at 6 months is -1.63.
3. Expected mean WLZ at 6 months is -1.23.
4. Expected mean weight gain in pregnancy is 7.55 kg (SD=3.23 kg).
5. Expected mean maternal weight at 6 m PP is 44.07 kg (SD=6.21 kg).

Stool Sub-Study: All substudy women in both groups will have stool collections at each indicated point in time. There are very few guidelines for sample size in microbiome studies. We consider these analyses to be exploratory and may provide important information regarding the mechanisms of how nutritional supplementation can improve birth outcomes and early infant growth.

Dietary Intake Sub-Study: We used two studies conducted among adults in the terai that use quantitative methods to estimate actual intake (Parajuli et al, 2012; Sudo et al, 2006). Both provided estimates of daily intake for a variety of nutrients for adult women and were very similar in their results. We used the average of their estimated intake of energy (kcal) and protein (g) and the associate average standard errors for our calculation. Mean energy intake was 1700 kcal/day (SD=350) and 42.3 g (SD=10.4) of protein. As this sub-study is designed to assess dietary diversion due to the supplement, we used a minimally detectable difference of -12% for energy and protein as an indicator that dietary diversion was occurring. Given these parameters, 120 persons per group will provide over 90% power for energy intake and approximately 85% power for protein intake.

Data Analysis, Phase 3: More detail will be available in the Statistical Analysis Plan document that will be posted to this site.

Data analysis will proceed in two phases, an exploratory data analysis phase followed by a confirmatory analysis phase and focuses on the specific aims of this project. The exploratory phase will involve final data cleaning and editing as well as examination of the distributions for all variables and the application of appropriate transformations. We will populate a CONSORT diagram. Next, comparisons will be made between the four treatment groups on a variety of variables at the household and individual levels to assess their comparability. All eligible birth outcomes will be limited to those measured within 72 hours of delivery.

Pregnancy Intervention Primary Aim: Data analysis will be by intent to treat. The proportion of babies born SGA (10th centile) will be compared in the two treatment groups using generalized estimating equations (GEE). An effect size will be estimated as the proportionate change in the intervention group relative to the control group. A 95% confidence interval will be calculated around this effect size estimate that accounts for the correlation within households. A secondary, post-hoc stratification by level of compliance with supplement use will be done within the active treatment group and the proportion SGA will be compared across groups. A dose-response effect will be estimated by linear regression techniques.

Secondary Aims 1, 2, and 3: A similar analysis to that of the primary aim will be done for the outcome ShGA (10th centile), SGA (3rd centile), and ShGA (3rd centile).

Secondary Aim 4: Mean birthweight and the distribution of birthweights will be compared by treatment group (supplementation during pregnancy versus not). Means and proportions below 2500 grams will be compared using GEE. A comparison of the full distribution of birthweights between treatment groups will also be done as previous research in this study area has indicated that treatment effects may vary by location on the birthweight distribution. (Katz et al, 2006; Dominici et al, 2006). A similar analysis of birth length will be conducted. A similar analysis will be conducted for the mean and distribution of gestational age and the proportion preterm (<37 weeks gestation).

Secondary Aim 5: Mean Length-for-Age, Weight-for-Age, Weight-for-Length, and proportions (<-2 Z scores) at 6 months of age will be compared by treatment group using GEE.

Post-Partum Intervention Primary Aim: Data analysis will be by intent to treat. The mean LAZ score among infants at 6 months of age will be compared in the two treatment groups using GEE. An effect size will be estimated as the proportionate change in the intervention group relative to the control group. A 95% confidence interval will be calculated around this effect size estimate that accounts for the correlation within clusters. A secondary, post-hoc stratification by level of compliance with supplement use during lactation will be done within the active treatment group and the mean LAZ score will be compared across groups. A dose-response effect will be estimated by linear regression techniques.

Secondary Aim 1: A similar analysis to that of the primary aim will be done for the outcome WAZ and WLZ scores.

Secondary Aim 2: Weight (and BMI) of mothers at 6 months post-partum will be compared by treatment group using GEE. An effect size will be estimated as the proportionate change in the intervention group relative to the control group. A 95% confidence interval will be calculated around this effect size estimate that accounts for the correlation within clusters. A secondary, post-hoc stratification by level of compliance with supplement use during lactation will be done within the active treatment group and the mean weight and BMI will be compared across groups. A dose-response effect will be estimated by linear regression techniques.

Combination of Pregnancy and Post-Partum Supplementation

Secondary Aim 1: The combined effect of both pregnancy and post-partum supplementation on 6 and 12 month LAZ, WAZ, and WLZ scores will be estimated two ways. First a stratified analysis will be done comparing mean and 95% CI on Z scores among control in both periods with pregnancy alone, post-partum alone, and both pregnancy and post-partum supplementation. For significance testing we have chosen the following 3 comparisons to apply tests of significance:

* Control in both periods versus post-partum alone.
* Pregnancy alone versus post-partum alone.
* Post-partum alone versus both pregnancy and post-partum. The second approach will be to model the effects of the treatment groups using linear regression models that include an interaction term for the combined treatment arm. A test of interaction will be used but we will primarily rely on interpreting the size of the interaction effect relative to the changes in the period-specific supplementation effects.

A variety of additional analyses will be conducted to explore the consistency of the main effects of these interventions.

Ethical Considerations The project has been approved by Institutional Review Boards (IRBs) at the George Washington University, the Johns Hopkins Bloomberg School of Public Health, and the Nepal Health Research Council. The IRB at the Harvard T.H. Chan School of Public Health has defered to the IRB of record at George Washington University.

Adverse Event Reporting Serious Adverse Events: Serious adverse events (SAE) under GCP guidelines include death, a life-threatening reaction to the supplement or other study procedure, hospitalization, significant or persistent disability or impairment, or a congenital anomaly/birth defect.

Other Adverse Events: These include any untoward medical event that occurs in a participant, any unfavorable sign or symptom of disease temporally associated with the provision of the supplement, or any noxious and unintended response to the supplement. Anticipated adverse events include signs/symptoms of allergic reaction to the supplement, preeclampsia, infection during pregnancy, gestational diabetes. Unanticipated adverse events are either unexpected in terms of nature, severity and frequency. An example would include newborn macrosomia (BW>97th centile according to InterGrowth21 standards).

All adverse events will be reported to the designated local investigator for review within 48 hours. If there is a possibility of the event being related to the study, a report will be made to the independent Safety Officer within 24 hours of receipt by the investigator. The Safety Officer will review the file and make a determination regarding attribution to study procedures or the intervention. If the adverse event is considered by the Safety Officer to be minor in severity, it will be logged and a summary of such events will be reported to the DSMB at their next meeting. If the severity of the adverse event is considered to be moderate or severe by the Safety Officer, he/she will indicate to the Principal Investigator that it should be reported to the DSMB and the cognizant IRBs immediately. The PI will then forward all materials together with the Safety Officer's summary to the DSMB and the IRBs.

ELIGIBILITY:
Inclusion Criteria:

* all women who become pregnant during an approximate 6-month period in two cohorts in a set of Nagarpalikas and Gaunpalikas in Sarlahi District, Nepal.

Exclusion Criteria:

* Women who do not intend to deliver their child in the study area.
* Women who are allergic to milk, nuts or soy.
* Women who are unwilling to commit to daily consumption of the nutritional supplement if they are randomized to an active treatment arm.
* Women who refuse to provide consent.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1944 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Small-for-Gestational-Age (<10th centile weight(g) for gestational age) | Within 72 hours of birth.
  The incidence of SGA (<10th centile) among live born infants whose birth weight(g) is measured within 72 hours of delivery. Comparison is between those supplemented during pregnancy versus those not.
Length-for-Age Z scores | 6 months of age
  Mean Length(cm)-for-age Z score among infants at 6 months of age. Comparison is between women supplemented during post-partum period versus those not.

SECONDARY OUTCOMES:
Short-for-Gestational-Age (<10th centile height(cm) for gestational age) | Within 72 hours of birth.
  The incidence of ShGA (<10th centile among live born infants whose birth length(cm) is measured within 72 hours of delivery.
Small-for-Gestational-Age (<3rd centile weight(g) for gestational age) | Within 72 hours of birth.
  The incidence of SGA (<3rd centile) among live born infants whose birth weight(g) is measured within 72 hours of delivery.
Short-for-Gestational-Age (<3rd centile height(cm) for gestational age) | Within 72 hours of birth.
  The incidence of ShGA (<3rd centile) among live born infants whose birth length(cm) is measured within 72 hours of delivery.
Birth weight | Within 72 hours of birth.
  Mean birthweight (g) among live born infants whose birthweight is measured within 72 hours of delivery.
Low birth weight (<2500 g) | Within 72 hours of birth.
  Proportion low birth weight (<2500 g) among live born infants whose birth weight is measured within 72 hours of delivery.
Birth Length | Within 72 hours of birth.
  Mean birth length (cm) among live born infants whose birth length is measured within 72 hours of delivery.
Gestational age | Birth
  Mean gestational age(weeks) among live born infants.
Proportion preterm (<37 weeks) | Birth
  Proportion preterm (<37 weeks gestation) among live born infants.
Prevalence of stunting | 6 and 12 months of age.
  Prevalence of Length(cm)-for-Age <-2 Z scores at 6 and 12 months of age among live born infants based on the WHO growth reference standards (WHO, 2006).
Weight-for-age | 6 & 12 months of age.
  Mean Weight(g)-for-Age Z score at 6 & 12 months of age among live born infants based on the WHO growth reference standards (WHO, 2006).
Prevalence of underweight | 6 & 12 months of age.
  Prevalence of Weight(g)-for-Age <-2 Z scores at 6 & 12 months of age among live born infants based on the WHO growth reference standards (WHO, 2006).
Weight-for-length | 6 & 12 months of age.
  Mean Weight(g)-for-Length(cm) Z score at 6 & 12 months of age among live born infants based on the WHO growth reference standards (WHO, 2006).
Prevalence of wasting | 6 & 12 months of age.
  Prevalence of Weight(g)-for-Length <-2 Z scores at 6 & 12 months of age among live born infants based on the WHO growth reference standards (WHO, 2006).
Maternal weight (kg). | Late pregnancy visit (~ 36 weeks) & 6 months post-partum.
  Mean maternal weight (kg) at late pregnancy visit (~ 36 weeks) & 6 months post-partum.
Maternal Body Mass Index (BMI) | Late pregnancy visit (~ 36 weeks) & 6 months post-partum.
  BMI (Weight(kg/Height(m)*2) at late pregnancy visit (~ 36 weeks) & 6 months post-postpartum
Microbiome Diversity - Mothers | Baseline enrollment, mid-2nd trimester, late pregnancy, 1-2 months post-partum, and 3-4 months post-partum
  PCR based measures of gut microbiome diversity during pregnancy and early lactation among women
Microbiome Diversity - Infants | 1-2 months of age and 3-4 months of age.
  PCR based measures of gut microbiome diversity among infants.
Gestational Weight Gain | From enrollment to the late pregnancy visit (34-36 weeks gestation).
  Change in maternal weight from enrollment to 36 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: James M Tielsch, PhD, Principal Investigator — George Washington University; Parul Christian, PhD, Principal Investigator — Johns Hopkins University; Tsering P Lama, PhD, Principal Investigator — Nepal Nutrition Intervention Project Sarlahi; Daniel Erchick, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Nepal Nutrition Intervention Project - Sarlahi, Hariaun, Sarlahi District, Nepal

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be available on a Gates Foundation supported website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months following article publication. No end date.
Access Criteria: Proposals should be directed to jtielsch@gwu.edu. To gain access, data requestors will need to sign a data access agreement. Data will be posted after 12 months to a website supported by the Bill and Melinda Gates Foundation.

REFERENCES:
- [Background] Bernard HR. Research methods in anthropology. 2nd ed. Thousand Oaks, CA: Sage Publications; 2006.
- [Background] Campbell RK, Talegawkar SA, Christian P, LeClerq SC, Khatry SK, Wu LS, West KP Jr. Seasonal dietary intakes and socioeconomic status among women in the Terai of Nepal. J Health Popul Nutr. 2014 Jun;32(2):198-216. PMID 25076658
- [Background] Constructing Grounded Theory: A practical guide through qualitative analysis Kathy Charmaz Constructing Grounded Theory: A practical guide through qualitative analysis Sage 224 pound19.99 0761973532 0761973532 [Formula: see text]. Nurse Res. 2006 Jul 1;13(4):84. doi: 10.7748/nr.13.4.84.s4. PMID 27702218
- [Background] Charmaz K. Constructing grounded theory: Sage; 2014.
- [Background] Christian P, Bunjun Srihari S, et al. Eating down in pregnancy: exploring food-related beliefs and practices of pregnancy in rural Nepal. Ecology of food and nutrition. 2006; 45(4):253-78.
- [Background] Consultants SR. Dedoose web application for managing, analyzing, and presenting qualitative and mixed methods research data. 7.0.23 ed. Los Angeles, CA: SocioCultural Research Consultants, LLC; 2016.
- [Background] de Graaf C, Kramer FM, Meiselman HL, Lesher LL, Baker-Fulco C, Hirsch ES, Warber J. Food acceptability in field studies with US army men and women: relationship with food intake and food choice after repeated exposures. Appetite. 2005 Feb;44(1):23-31. doi: 10.1016/j.appet.2004.08.008. Epub 2004 Nov 13. PMID 15604031
- [Background] Dominici F, Zeger SL, Parmigiani G, et al. Estimating percentile-specific effects: a case study of micronutrient supplementation, birth weight, and infant mortality. J R Stat Soc Ser C Appl Stat. 2006; 50:1-20.
- [Background] Duggan C, Srinivasan K, Thomas T, Samuel T, Rajendran R, Muthayya S, Finkelstein JL, Lukose A, Fawzi W, Allen LH, Bosch RJ, Kurpad AV. Vitamin B-12 supplementation during pregnancy and early lactation increases maternal, breast milk, and infant measures of vitamin B-12 status. J Nutr. 2014 May;144(5):758-64. doi: 10.3945/jn.113.187278. Epub 2014 Mar 5. PMID 24598885
- [Background] Expert Consultation held at The Bill and Melinda Gates Foundation. Framework and specifications for the nutritional composition of a food supplement for pregnant and lactating women (PLW) in undernourished and low income settings. Bill and Melinda Gates Foundation, 2016 Sept 19-20, Seattle, WA.
- [Background] Furuta M, Salway S. Women's position within the household as a determinant of maternal health care use in Nepal. Int Fam Plan Perspect. 2006 Mar;32(1):17-27. doi: 10.1363/3201706. PMID 16723298
- [Background] Glesne C, Peshkin A. Becoming qualitative researchers: an introduction. White Plains, NY: Longman; 1992.
- [Background] Gittelsohn J. Opening the box: intrahousehold food allocation in rural Nepal. Soc Sci Med. 1991;33(10):1141-54. doi: 10.1016/0277-9536(91)90230-a. PMID 1767284
- [Background] Gittelsohn J, Thapa M, Landman LT. Cultural factors, caloric intake and micronutrient sufficiency in rural Nepali households. Soc Sci Med. 1997 Jun;44(11):1739-49. doi: 10.1016/s0277-9536(96)00375-9. PMID 9178416
- [Background] Haider BA, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2017 Apr 13;4(4):CD004905. doi: 10.1002/14651858.CD004905.pub5. PMID 28407219
- [Background] Hampel D, Shahab-Ferdows S, Islam MM, Peerson JM, Allen LH. Vitamin Concentrations in Human Milk Vary with Time within Feed, Circadian Rhythm, and Single-Dose Supplementation. J Nutr. 2017 Apr;147(4):603-611. doi: 10.3945/jn.116.242941. Epub 2017 Feb 15. PMID 28202638
- [Background] Hayes RJ, Moulton LH. Cluster Randomized Trials. Boca Raton FL: Chapman & Hall/CRC, 2009.
- [Background] Henjum S, Torheim LE, Thorne-Lyman AL, Chandyo R, Fawzi WW, Shrestha PS, Strand TA. Low dietary diversity and micronutrient adequacy among lactating women in a peri-urban area of Nepal. Public Health Nutr. 2015 Dec;18(17):3201-10. doi: 10.1017/S1368980015000671. Epub 2015 Mar 31. PMID 25824344
- [Background] Henjum S, Lie O, Ulak M, Thorne-Lyman AL, Chandyo RK, Shrestha PS, W Fawzi W, Strand TA, Kjellevold M. Erythrocyte fatty acid composition of Nepal breast-fed infants. Eur J Nutr. 2018 Apr;57(3):1003-1013. doi: 10.1007/s00394-017-1384-4. Epub 2017 Feb 25. PMID 28238109
- [Background] Imdad A, Bhutta ZA. Maternal nutrition and birth outcomes: effect of balanced protein-energy supplementation. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:178-90. doi: 10.1111/j.1365-3016.2012.01308.x. PMID 22742610
- [Background] Janmohamed A, Karakochuk CD, Boungnasiri S, Chapman GE, Janssen PA, Brant R, Green TJ, McLean J. Prenatal supplementation with Corn Soya Blend Plus reduces the risk of maternal anemia in late gestation and lowers the rate of preterm birth but does not significantly improve maternal weight gain and birth anthropometric measurements in rural Cambodian women: a randomized trial. Am J Clin Nutr. 2016 Feb;103(2):559-66. doi: 10.3945/ajcn.114.104034. Epub 2016 Jan 6. PMID 26739037
- [Background] Jiang T, Christian P, Khatry SK, Wu L, West KP Jr. Micronutrient deficiencies in early pregnancy are common, concurrent, and vary by season among rural Nepali pregnant women. J Nutr. 2005 May;135(5):1106-12. doi: 10.1093/jn/135.5.1106. PMID 15867289
- [Background] Jones KM, Specio SE, Shrestha P, Brown KH, Allen LH. Nutrition knowledge and practices, and consumption of vitamin A--rich plants by rural Nepali participants and nonparticipants in a kitchen-garden program. Food Nutr Bull. 2005 Jun;26(2):198-208. doi: 10.1177/156482650502600204. PMID 16060221
- [Background] Katz J, Christian P, Dominici F, Zeger SL. Treatment effects of maternal micronutrient supplementation vary by percentiles of the birth weight distribution in rural Nepal. J Nutr. 2006 May;136(5):1389-94. doi: 10.1093/jn/136.5.1389. PMID 16614435
- [Background] Kodish S, Aburto N, Hambayi MN, Kennedy C, Gittelsohn J. Identifying the Sociocultural Barriers and Facilitating Factors to Nutrition-related Behavior Change: Formative Research for a Stunting Prevention Program in Ntchisi, Malawi. Food Nutr Bull. 2015 Jun;36(2):138-53. doi: 10.1177/0379572115586784. PMID 26121699
- [Background] Kozuki N, Lee AC, Black RE, Katz J. Nutritional and Reproductive Risk Factors for Small for Gestational Age and Preterm Births. Nestle Nutr Inst Workshop Ser. 2015;81:17-28. doi: 10.1159/000365799. Epub 2015 Jun 16. PMID 26111560
- [Background] Lawless HT, Heymann H. Sensory evaluation of food: principles and practices. 2nd ed. New York: Springer; 2010. xxiii, 596 p. p.
- [Background] Manandhar DS, Osrin D, Shrestha BP, Mesko N, Morrison J, Tumbahangphe KM, Tamang S, Thapa S, Shrestha D, Thapa B, Shrestha JR, Wade A, Borghi J, Standing H, Manandhar M, Costello AM; Members of the MIRA Makwanpur trial team. Effect of a participatory intervention with women's groups on birth outcomes in Nepal: cluster-randomised controlled trial. Lancet. 2004 Sep 11-17;364(9438):970-9. doi: 10.1016/S0140-6736(04)17021-9. PMID 15364188
- [Background] Ministry of Health, Nepal; New ERA; and ICF. 2017. Nepal Demographic and Health Survey 2016: Key Indicators. Kathmandu, Nepal: Ministry of Health, Nepal.
- [Background] Ota E, Hori H, Mori R, Tobe-Gai R, Farrar D. Antenatal dietary education and supplementation to increase energy and protein intake. Cochrane Database Syst Rev. 2015 Jun 2;2015(6):CD000032. doi: 10.1002/14651858.CD000032.pub3. PMID 26031211
- [Background] Parajuli RP, Umezaki M, Watanabe C. Diet among people in the Terai region of Nepal, an area of micronutrient deficiency. J Biosoc Sci. 2012 Jul;44(4):401-15. doi: 10.1017/S0021932012000065. Epub 2012 Mar 19. PMID 22424573
- [Background] Rahman MM, Abe SK, Kanda M, Narita S, Rahman MS, Bilano V, Ota E, Gilmour S, Shibuya K. Maternal body mass index and risk of birth and maternal health outcomes in low- and middle-income countries: a systematic review and meta-analysis. Obes Rev. 2015 Sep;16(9):758-70. doi: 10.1111/obr.12293. Epub 2015 Jun 11. PMID 26094567
- [Background] Ridder HG, Miles MB, Huberman AM, Saldana J. Qualitative data analysis: a methods source book. 3rds ed. Thousand Oaks, CA: Sage Publications; 2014.
- [Background] Sandelowski M. Combining qualitative and quantitative sampling, data collection, and analysis techniques in mixed-method studies. Res Nurs Health. 2000 Jun;23(3):246-55. doi: 10.1002/1098-240x(200006)23:33.0.co;2-h. PMID 10871540
- [Background] Simkhada B, Porter MA, van Teijlingen ER. The role of mothers-in-law in antenatal care decision-making in Nepal: a qualitative study. BMC Pregnancy Childbirth. 2010 Jul 1;10:34. doi: 10.1186/1471-2393-10-34. PMID 20594340
- [Background] Stevens B, Buettner P, Watt K, Clough A, Brimblecombe J, Judd J. The effect of balanced protein energy supplementation in undernourished pregnant women and child physical growth in low- and middle-income countries: a systematic review and meta-analysis. Matern Child Nutr. 2015 Oct;11(4):415-32. doi: 10.1111/mcn.12183. Epub 2015 Apr 7. PMID 25857334
- [Background] Sudo N, Sekiyama M, Maharjan M, Ohtsuka R. Gender differences in dietary intake among adults of Hindu communities in lowland Nepal: assessment of portion sizes and food consumption frequencies. Eur J Clin Nutr. 2006 Apr;60(4):469-77. doi: 10.1038/sj.ejcn.1602339. PMID 16391580
- [Background] Department of Homeland Security; Department of Agriculture; Department of Energy; National Aeronautics and Space Administration; Department of Commerce; Social Security Administration; Agency for International Development; Department of Housing and Urban Development; Department of Labor; Department of Defense; Department of Education; Department of Veterans Affairs; Environmental Protection Agency; Department of Health and Human Services; National Science Foundation; Department of Transportation. Federal Policy for the Protection of Human Subjects. Final rule. Fed Regist. 2017 Jan 19;82(12):7149-274. PMID 28106360
- [Background] Villar J, Cheikh Ismail L, Victora CG, Ohuma EO, Bertino E, Altman DG, Lambert A, Papageorghiou AT, Carvalho M, Jaffer YA, Gravett MG, Purwar M, Frederick IO, Noble AJ, Pang R, Barros FC, Chumlea C, Bhutta ZA, Kennedy SH; International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st). International standards for newborn weight, length, and head circumference by gestational age and sex: the Newborn Cross-Sectional Study of the INTERGROWTH-21st Project. Lancet. 2014 Sep 6;384(9946):857-68. doi: 10.1016/S0140-6736(14)60932-6. PMID 25209487
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] WHO. Handbook for Good Clincial Research Practice (GCP): Guidance for Implementation. World Health Organization, Geneva, 2005.
- [Background] World Health Organization. WHO Child Growth Standards: Methods and development: Length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age: methods and development. World Health Organization, Geneva, 2006.
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Derived] Erchick DJ, Lama TP, Khatry SK, Katz J, Mullany LC, Zavala E, LeClerq SC, Christian P, Tielsch JM. Supplementation with fortified balanced energy-protein during pregnancy and lactation and its effects on birth outcomes and infant growth in southern Nepal: protocol of a 2x2 factorial randomised trial. BMJ Paediatr Open. 2023 Nov;7(1):e002229. doi: 10.1136/bmjpo-2023-002229. PMID 37923345